CLINICAL TRIAL: NCT05586724
Title: Safety of Oral Micronized Progesterone Versus Norethisterone Acetate in Continuous Combination With Oral Estrogen as Menopausal Hormone Therapy - a Double-blind Randomized Study- PROBES Study (Progesterone Breast Endometrial Safety Study)
Brief Title: Micronized Progesterone Versus Norethisterone Acetate in Combination With Estrogen as Menopausal Hormone Therapy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Angelica Lindén Hirschberg (Other)
Responsible Party: Sponsor-Investigator, Angelica Lindén Hirschberg, Professor, MD, PhD, Karolinska University Hospital
Organization: Karolinska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2021-001624-17
Record Dates: First submitted 2022-10-09; First posted 2022-10-19 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Menopausal Symptoms
Keywords: Menopausal hormone therapy; Climacteric symptoms; Progesterone; Progestogens; Breast safety; Endometrial safety
MeSH Terms: interventions — Progesterone; Estrogens; Norethindrone Acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Micronized progesterone in continuous combination with oral estrogen (Active Comparator): Capsule 100 mg mP (Utrogestan®) orally per day in continuous combination with 1 mg encapsulated estradiol (Estrofem®)
  Interventions: Drug: Micronized progesterone in continuous combination with oral estrogen
- Norethisterone acetate in continuous combination with oral estrogen (Active Comparator): Capsule 0.5 mg NETA/ 1 mg estradiol (Activelle®) orally per day (encapsulated and identical to Estrofem® and one matched placebo to Utrogestan.
  Interventions: Drug: Norethisterone acetate in continuous combination with oral estrogen

INTERVENTIONS:
Drug: Micronized progesterone in continuous combination with oral estrogen — Capsule 100 mg mP (Utrogestan®) orally per day in continuous combination with 1 mg encapsulated estradiol (Estrofem®)
  Arms: Micronized progesterone in continuous combination with oral estrogen
Drug: Norethisterone acetate in continuous combination with oral estrogen — Capsule 0.5 mg NETA/ 1 mg estradiol (Activelle®) orally per day (encapsulated and identical to Estrofem® and one matched placebo to Utrogestan
  Arms: Norethisterone acetate in continuous combination with oral estrogen

SUMMARY:
About one third of all women during menopausal transition have significant climacteric symptoms with considerable impact on quality of life. Meta-analysis has shown a beneficial risk profile with menopausal hormone therapy (MHT) for women 50 to 60 years. Still, there is a great need to find safe MHT able to control excessive endometrial stimulation by estrogen without stimulatory effects on the breast by the combination of estrogen/progestogen. Recent observational studies indicate a lower risk for breast cancer using micronized progesterone (mP) combined with estrogen but increased risk of endometrial cancer than by standard MHT. In a randomized trial, the balance between benefits and risks of mP vs. progestogens (norethisterone (NETA)) in combination with estrogen will be explored. For apparent reasons, long-term largescale clinical trials with endometrial and breast cancer as the primary endpoints, are not feasible. However, much knowledge can be obtained using relevant surrogate markers. Mammographic breast density is a strong risk factor for breast cancer, and endometrial hyperplasia is a strong risk factor for endometrial cancer. The primary objective is to compare the effects of one year treatment with mP versus progestogen, in combination with estradiol on mammographic breast density. Furthermore, to evaluate the effect of one year treatment with mP in continuous combination with estradiol on endometrial pathology (hyperplasia and cancer).

DETAILED DESCRIPTION:
Postmenopausal women with climacteric symptoms will be randomized (1:1) to double blind treatment with oral mP or NETA in combination with oral estradiol. For the breast part, a power analysis revealed that 91 women/group would be sufficient to detect a significant difference in mammographic breast density between the groups at the 5%-level (two-sided) with 80% power. Considering the estimated rate of discontinuation and incomplete data, the target sample for the breast part is 260 patients. For the endometrial part, it is estimated that two or less women with serious adverse endometrial outcomes would result in an annual incidence of endometrial pathology of 0.67% or less with an upper bound of the one-sided 95% CI of 2.08% or less. Considering the estimated rate of discontinuation and incomplete data in the mP + estradiol group, the target sample for this part of the study is 390 patients. The total number of patients in part 1 and 2 will be 520.

Mammography at baseline and after 12 months of treatment will be assessed by independent radiologists at the Karolinska University Hospital blinded to treatment. In addition to visual judgment, a computer based quantitative assessment will be performed. All mammograms will be anonymous so that the operator will be unaware of the patient's identity and type of treatment. Percentage change in mammographic density will be evaluated and compared between the groups.

Endometrial biopsies at baseline and after 12 months of treatment will be evaluated by two independent pathologists at the Karolinska University Hospital for the incidence of endometrial pathology (hyperplasia or cancer) in the mP + estradiol group. Furthermore, immunostaining of the proliferation marker Ki-67, and other markers related to proliferation and apoptosis will be analyzed and compared between groups.

Different validated self-assessment questionnaires will be used for screening of mood disorders like depression and anxiety, as well as quality of life and menopausal symptoms. The Patient Health Questionnaire (PHQ-9) is a tool for screening, diagnosing, and measuring the severity of depression. The Hospital Anxiety and Depression Scale (HADS) is an instrument for detecting states of depression and anxiety in the setting of a hospital or medical outpatient clinic. Health related quality of life is measured using the Psychological General Well-Being Index (PGWB). The Women's Health Questionnaire (WHQ) measures menopausal symptoms. The change in scores will be compared between the groups.

Blood lipid profile, serum hormones, growth and metabolic factors, and coagulation factors will be analyzed.

The gut- and vaginal microbiome will be characterized and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Healthy and naturally postmenopausal women (more than one year since last menstruation or FSH > 40 IE/L) with climacteric symptoms (sweating, hot flush and/or sleep problems) that adversely affect the quality of life
* Age 45-60 years
* BMI > 19 kg/m2 and ≤ 32 kg/m2
* Intact uterus
* In case of previous MHT use, washout 8 weeks for oral MHT and 4 weeks for transdermal MHT or local estrogen treatment before screening
* Written informed consent

Exclusion Criteria:

* Previous history or risk factors for breast cancer, breast cancer in situ or abnormal mammogram at baseline as assessed clinically by a radiology expert
* Previous history or risk factors for endometrial cancer or hyperplasia or abnormal/proliferative endometrial biopsy at baseline
* Vaginal bleeding
* Any concomitant medical treatment except for well-controlled hypertension, non-insulin treated type 2 diabetes, asthma and hypothyroidism
* History or presence of or risk factor for cardiovascular disease including thromboembolic disorder or cerebrovascular disease
* History or presence of liver and gallbladder disease, familial hyperlipidemia, epilepsy or classical migraine with aura
* History or presence of clinically significant depression or other psychiatric disorder that might in anyway compromise the performance of the trial or undermine its scientific validity
* Porphyria, Systemic lupus erythematosus and otosclerosis
* Current use of MHT or local estrogen treatment
* Alcohol and/or drug abuse
* Clinically significant findings on physical and/or gynecological examination at baseline
* Hypersensitivity to any of the study treatments

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 520 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Mammographic breast density | At baseline and 12 months treatment
  Percentage change in mammographic density
Endometrial pathology | At baseline and 12 months treatment
  The incidence of endometrial pathology (hyperplasia or cancer)

SECONDARY OUTCOMES:
Breast cell proliferation | At baseline and 12 months treatment
  Percentage change in breast cell proliferation (proliferation marker Ki-67)
Endometrial histology and cell proliferation | At baseline and 12 months treatment
  Percentage change in endometrial cell proliferation (histology classification and proliferation marker Ki-67)
Endometrial thickness | At baseline and 12 months treatment
  Change in endometrial thickness by ultrasound
Bleeding pattern | 3, 6, 9 and 12 months
  Bleeding patterns registered in diary (number of days of bleedings)
Gene and protein expression of growth factors and apoptosis markers in breast and endometrial tissue | At baseline and 12 months treatment
  Change in gene and protein expression (proliferation and apoptosis markers)
Depression (PHQ-9) | At baseline and 12 months treatment
  Change in score of PHQ-9: A 4-point scale where a larger value reflects more depression.
Anxiety (HADS) | At baseline and 12 months treatment
  Change in score of HADS: A 4-point scale where a larger value reflects more anxiety.
Quality of life (PGWB) | At baseline and 12 months treatment
  Change in score of PGWBI, where a where a higher score reflects more well-being.
Menopausal symptoms (WHQ) | At baseline and 12 months treatment
  WHQ: A 4-point scale where a larger value reflects less menopausal symptoms.
Serum levels of hormones, growth factors, lipids and coagulation factors. | At baseline and 12 months treatment
  Change in serum levels of these markers
Gut- and vaginal microbiome | At baseline and 12 months treatment
  Change in microbiome diversity and relative abundance of different microbial species.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be available to external researchers upon reasonable request after publication of the results and approval of the study management team.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Earliest from January 2028 and for ten years ahead.
Access Criteria: Investigators whose proposed use of the data has been approved by the study management team.
  To achieve aims in the approved proposal.
  Proposals should be directed to angelica.hirschberg.linden@ki.se. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Bofill Rodriguez M, Yong LN, Mirkov S, Bekos C, Lethaby A, Farquhar C. Long-term hormone therapy for perimenopausal and postmenopausal women. Cochrane Database Syst Rev. 2025 Nov 27;11(11):CD004143. doi: 10.1002/14651858.CD004143.pub6. PMID 41307293
- [Derived] Lundell C, Stergiopoulos N, Blomberg L, Ujvari D, Schuppe-Koistinen I, Kopp-Kallner H, Iliadis SI, Skalkidou A, Hirschberg AL. Breast and endometrial safety of micronised progesterone versus norethisterone acetate in menopausal hormone therapy (PROBES): study protocol of a double-blind randomised controlled trial. BMJ Open. 2024 Oct 23;14(10):e082749. doi: 10.1136/bmjopen-2023-082749. PMID 39448218